CLINICAL TRIAL: NCT03896958
Title: The PIONEER Initiative: Precision Insights On N-of-1 Effectiveness Research. Tissue Ownership by the Individual With the Return of Actionable Information to the Individual Patient and Physician (Precision Oncology)
Brief Title: The PIONEER Initiative: Precision Insights On N-of-1 Ex Vivo Effectiveness Research Based on Individual Tumor Ownership (Precision Oncology)
Acronym: PIONEER
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: SpeciCare (Industry)
Collaborators: Georgia Institute of Technology (Other); Predictive Oncology (Unknown); University of Washington (Other); Netnoids (Unknown); Northeast Georgia Hospital System (Unknown)
Responsible Party: Sponsor
Other Study IDs: MYCT001
Record Dates: First submitted 2019-03-26; First posted 2019-04-01 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Cancer, All Types; Cancer of Liver; Cancer of Stomach; Cancer of Head and Neck; Cancer of Rectum; Cancer of Kidney; Cancer of Esophagus; Cancer of Colon; Cancer Skin; Cancer of Cervix; Cancer, Metastatic; Cancer of Larynx; Cancer of Neck; Cancer of Lung; Cancer of Brain and Nervous System; Cancer of Vulva, Disseminated; Cancer of Pancreas; Sarcoma; GIST; Small-cell Lung Cancer; Adenocarcinoma Lung; Cancer of Prostate; Cancer, Advanced; Adrenal Cancer; Testicular Cancer; Uterine Cancer; Bronchoalveolar Cell Lung Cancer; Cancer Unknown Primary; Glioblastoma Multiforme; Oligodendroglioma; Breast Cancer; Renal Cell Carcinoma; Hepatocellular Carcinoma; Cholangiocarcinoma; Squamous Cell Carcinoma; Transitional Cell Carcinoma; Cancer, Other; Cancer, Anal; Melanoma; Cancer, Bile Duct; Cancer, Bladder; Cancer Cords Vocal; Cancers Cell Neuroendocrine; Cancer Differentiated Poorly; Cancer, Anaplastic Thyroid
MeSH Terms: conditions — Neoplasms; Liver Neoplasms; Stomach Neoplasms; Head and Neck Neoplasms; Rectal Neoplasms; Kidney Neoplasms; Esophageal Neoplasms; Colonic Neoplasms; Skin Neoplasms; Uterine Cervical Neoplasms; Neoplasm Metastasis; Laryngeal Neoplasms; Lung Neoplasms; Brain Neoplasms; Neurologic Manifestations; Vulvar Neoplasms; Pancreatic Neoplasms; Sarcoma; Small Cell Lung Carcinoma; Adenocarcinoma of Lung; Prostatic Neoplasms; Adrenal Gland Neoplasms; Testicular Neoplasms; Uterine Neoplasms; Adenocarcinoma, Bronchiolo-Alveolar; Neoplasms, Unknown Primary; Glioblastoma; Oligodendroglioma; Breast Neoplasms; Carcinoma, Renal Cell; Carcinoma, Hepatocellular; Cholangiocarcinoma; Carcinoma, Squamous Cell; Carcinoma, Transitional Cell; Anus Neoplasms; Melanoma; Bile Duct Neoplasms; Urinary Bladder Neoplasms; Thyroid Carcinoma, Anaplastic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biospecimens are saved in fresh and cryopreserved state. Also, FFPE, DNA, and RNA extraction.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The PIONEER Initiative stands for Precision Insights On N-of-1 Ex vivo Effectiveness Research. The PIONEER Initiative is designed to provide access to functional precision medicine to any cancer patient with any tumor at any medical facility. Tumor tissue is saved at time of biopsy or surgery in multiple formats, including fresh and cryopreserved as a living biospecimen. SpeciCare assists with access to clinical records in order to provide information back to the patient and the patient's clinical care team. The biospecimen tumor tissue is stored in a bio-storage facility and can be shipped anywhere the patient and the clinical team require for further testing. Additionally, the cryopreservation of the biospecimen allows for decisions about testing to be made at a later date. It also facilitates participation in clinical trials. The ability to return research information from this repository back to the patient is the primary end point of the study. The secondary end point is the subjective assessment by the patient and his or her physician as to the potential benefit that this additional information provides over standard of care. Overall the goal of PIONEER is to enable best in class functional precision testing of a patient's tumor tissue to help guide optimal therapy (to date this type of analysis includes organoid drug screening approaches in addition to traditional genomic profiling).

DETAILED DESCRIPTION:
The PIONEER Initiative is a lead clinical trial designed to provide the foundation for subsequent adaptive trials. The mission with this and subsequent trial activity will be to demonstrate the utility of carrying out functional precision medicine in that cohort of patients who receive local cancer care at institutions that do not have significant research capabilities or are not NCI-designated cancer centers. As discussed above, the vast majority of cancer patients (~85%) are in this category. It is imperative to open up the possibility of best-in-class functional precision medicine testing to these patients. Core aspects of the PIONEER Initiative include recruiting a cadre of up to 200 patients, showing that proof of concept in a more limited set of patients can ultimately scale to arbitrarily large numbers of patients. It is anticipated that PIONEER will continue as the foundation for subsequent clinical trials into the indefinite future. This evolving trial structure fills an important unmet need within the broader cancer community since the primary mission is the return of actionable information in order to positively impact care.

The underlying basic assumption of the PIONEER Initiative is that the ability to receive the best in cancer care should not be restricted as to location, age, or medical condition. The PIONEER Initiative design facilitates inclusion of subjects across all these divides, thus providing beneficence to all participants. A key aspect of the PIONEER Initiative is to provide patient benefit through a data and tissue biorepository to be utilized by researchers to discover new cancer diagnostics, treatment therapies and preventive strategies. Additionally, the data and samples will be used to improve existing treatments and to understand, at the molecular level, changes occurring during transition from illness to remission and/or relapse. SpeciCare, through the PIONEER Initiative, will store de-identified self-reported data, medical records, and biological samples from individuals who consent to participate in PIONEER. PIONEER will obtain further study and testing as appropriate and return results, through CLIA certified labs, through research vetted by CLIA testing, and, as enabled by current regulatory standards, through delivery of research results back to the patient and patient's clinical care team.

SPECIFIC OBJECTIVES

1. To establish a data and tissue biobank comprised of high quality biological specimens and associated clinical data that will support drug discovery, diagnostic assay development, oncology biomarker discovery, molecular biology, immuno-oncology therapies, translational medicine and other future discoveries as novel methods become available.
2. To facilitate and accelerate oncology research, including genetic research (e.g. whole genome sequencing), by providing a pipeline of high quality specimens and associated clinical data for researchers to access.

ELIGIBILITY:
Inclusion Criteria:

- All patients diagnosed with cancer and all patients at risk of cancer

Exclusion Criteria:

-Patients who decline definitive therapies Patients with comorbidities that prevent definitive therapies Patients on hospice

Ages: 1 Month to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The primary target study group is all patients with a cancer serious enough to put the patient at risk of morbidity or death.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-03-21 (Actual); Primary Completion 2024-03-12 (Estimated); Study Completion 2024-03-12 (Estimated)

PRIMARY OUTCOMES:
Return of research information | Two Years
  Monitor the ability to return research and study information back to the individual patient and cancer care team over time. We will calculate the % of patients that carry out additional genomic testing, % of patients that carry out additional functional precision testing, and % of clinicians that report that they altered their clinical therapeutic regiments based upon these results
Assessment of benefit of return of research results | Two Years
  Survey of study subjects and physicians as to the benefit or not of access to this additional data in attempting to improve upon standard of care of the day. We will calculate this as a % of patients.
Assessment of benefit of return of research results by SpeciCare Outcome Monitor Board | Two Years
  The primary mission of our team is to assess benefit of patient tissue ownership and functional testing to the standard of care process. We will calculate this as a % of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Ken Dixon, MD, Principal Investigator — SpeciCare
Locations (1):
- Specicare, Gainesville, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with strategic partners with appropriate IRB vetting.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Within six months of completion of study and/or publication of data driven by the study.
Access Criteria: SpeciCare has a data access committee, to which researchers can apply and receive data pending approval of this committee.